CLINICAL TRIAL: NCT04280627
Title: Changes in the Microbiome Associated With Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: B00150
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Microbiota
Keywords: microbiome
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will involve the collection of oral swabs, saliva, urine and faeces samples, blood and skin scrapings from 50 patients (phase 1) and up to 300 patients (phase 2) before (day of arrival in hospital day 0 and after kidney and pancreas transplantation day 1, week 1, 3, 6,12 months.
  In addition duodenal fluid from the donor duodenum which is opened at the time of pancreas transplantation will also be taken in theatre for analysis.
  Similar samples will be obtained from deceased multi-organ donors who have consent for research.
  Similar samples will also be taken from living kidney donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample Collection — This study will involve the collection of oral swabs, saliva, urine and faeces samples, blood and skin scrapings from patients before and after kidney and pancreas transplantation at day 0, day 1, week 1 and at 3, 6 and 12 months post-transplant.

SUMMARY:
To study the effects of organ transplantation and immunosuppression on the human microbiome, and to understand the interlinkage of changes in the microbiome with clinical events surrounding transplantation, and graft and patient clinical outcomes.

DETAILED DESCRIPTION:
This study will involve the collection of oral swabs, saliva, urine and rectal swabs, blood and skin scrapings from patients before and after kidney and pancreas transplantation. At Day 0 and day 1, week 1, and at 3, 6, and 12 months.

These samples will be collected longitudinally over a period of one year after transplantation and will be analysed using 16s rRNA gene sequencing in order to capture the dynamics of the microbiome after exposure to surgery, immunosuppression and the specific medication necessary during the process of transplantation.

Two groups of recipients will be recruited, the first one includes kidney and/or pancreas transplant recipients from both deceased and living donors.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Under 75 years
* Participants must be able to receive and understand English verbal and written information regarding the study and give written, informed consent.
* Participants will be recipients of pancreas or kidney allografts

Exclusion Criteria:

* Outside of stated age range.
* Unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney and Transplant Recipients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Microbiome following transplantation | 3 years
  The tissue samples will be examined to identify any microbial organisms. This process will involve cell identification and quantification using standard biological markers to identify cell types and numbers

CONTACTS AND LOCATIONS:
Overall Officials: Titus Augustine, FRCP, Principal Investigator — Consultant Transplant Surgeon; Oana Piscoran, MD, Principal Investigator — Clinical Research Fellow
Locations (1):
- Manchester University NHS Foundationn Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No